CLINICAL TRIAL: NCT03840785
Title: Effect of Argentine Tango Protocol on Total Physical Activity in Patients With Chronic Inflammatory Arthritis
Brief Title: Inflammatory Arthritis and Tango
Acronym: IATANGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHU-422; 2018-A01563-52 (Other: 2018-A01563-52)
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Rheumatoid Arthritis (RA); Spondyloarthritis (SA)
Keywords: Chronic inflammatory arthritis; argentine tango; physical activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Motor Activity

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group A (Experimental): 2 tango session per week during 6 month (M0 to M6)
  Interventions: Other: Argentine tango
- Control group B (Placebo Comparator): 2 tango session per week during 3 month (M3 to M6)
  Interventions: Other: Argentine tango

INTERVENTIONS:
Other: Argentine tango — Argentine tango sessions will consist of:
  * Body perception and body control: sitting, standing then moving around four axes : space, time, energy, gravity.
  * Awareness of oneself, of other and music: listening, communication, touch, empathy, kinesthesia, letting go, feeling

SUMMARY:
The hypothesis is that pleasure brought by argentine tango practice would increase total physical activity of patients with chronic inflammatory arthritis.

DETAILED DESCRIPTION:
Selection and inclusion of patients will be done by principal investigator of Rheumatology Department. After verification of inclusion and non-inclusion criteria by principal investigator and signature of consent, patients will be randomized by 1: 1 randomization (centralized randomization by statistician into 2 groups at M0). They will participate in sessions in a deferred manner due to two per week for each group:

* Interventional "A" group: 48 sessions (on average 2/week) performed from M0 to M6 in 30 patients.
* Control "B" group: 24 sessions (on average 2/week) performed from M3 to M6 in 30 patients.

Patients of "B" group will be not performing sessions with "A" group patients. Sessions lasting about 60 minutes will be proposed from Monday to Friday in a room planned from this activity within the CHU. They will be adapted and personalized according to each one. Evaluations will be carried out for group 1 (interventional) before the first session of tango at M0, before the session at M3 and at the end of the protocol at M6. The same evaluations will be carried out for group B (control) at M0, before first session of tango at M3 and at the end of the protocol.

Assessment of pain and stress will be done before and after each session. Final assessment will be done at 6 months after randomization. Fitness assessment and tango sessions will be conducted by an argentine tango teacher

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old with RA (ACR/EULAR criteria) in remission (CDAI ≤2.8) or with low disease activity (CDAI ≤10), or with SA (ASAS criteria) with activity deemed stable by rheumatologist.
* Patient able to walk without help
* Patient able to complete a questionnaire
* Patient giving informed consent.
* Patient covered by social security

Exclusion Criteria:

* Patient with disorder of higher mental function or psychiatric disorders.
* Patient practicing argentine tango.
* Patient with an absolute contraindication to physical activity.
* Protected populations: pregnant women, breastfeeding women, tutorship, trusteeship, deprived of liberty, safeguard of justice.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change in total physical activity time | between month 0 and month3
  Total physical activity measured by Modified Global Physical Activity Questionnaire (GPAQ) between M0 and M3. Modified Global Physical Activity Questionnaire (GPAQ) questionnaire provides information on the time spent on different activities: work activity, utilitarian travel, hobbies and home-based activities. A specific energy expenditure is associated with each physical activity, which makes it possible to estimate the overall energy expenditure of the patients. It also provides information on sedentary time.

SECONDARY OUTCOMES:
Change in total physical activity time | at 3 months and 6 months
  Recording of total physical activity over a week by an accelerometer worn at the waist
Physical activity time of light intensity | at 3 months and 6 months
  measured by an accelerometer and measured by the modified GPAQ questionnaire (Global Physical Activity Questionnaire).Global Physical Activity Questionnaire (GPAQ) provides information on the time spent on different activities: work activity, utilitarian travel, hobbies and home-based activities.
Physical activity time of moderate intensit | at 3 months and 6 months
  measured by an accelerometer and measured by the modified GPAQ questionnaire (Global Physical Activity Questionnaire). Global Physical Activity Questionnaire (GPAQ) provides information on the time spent on different activities: work activity, utilitarian travel, hobbies and home-based activities.
Physical activity time of high intensity | at 3 months and 6 months
  : measured by an accelerometer and measured by the modified GPAQ. Global Physical Activity Questionnaire (GPAQ) provides information on the time spent on different activities: work activity, utilitarian travel, hobbies and home-based activities. questionnaire (Global Physical Activity Questionnaire)
Sedentary time by the modified GPAQ questionnaire (Global Physical Activity)Questionnaire) | at 3 months and 6 months
  Recording sedentary time over a week by an accelerometer worn at the waist

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Biswas A, Oh PI, Faulkner GE, Bajaj RR, Silver MA, Mitchell MS, Alter DA. Sedentary time and its association with risk for disease incidence, mortality, and hospitalization in adults: a systematic review and meta-analysis. Ann Intern Med. 2015 Jan 20;162(2):123-32. doi: 10.7326/M14-1651. PMID 25599350
- [Background] Sokka T, Hakkinen A. Poor physical fitness and performance as predictors of mortality in normal populations and patients with rheumatic and other diseases. Clin Exp Rheumatol. 2008 Sep-Oct;26(5 Suppl 51):S14-20. PMID 19026141
- [Background] Garner S, Fenton T, Martin L, Creaser C, Johns C, Barnabe C. Personalized diet and exercise recommendations in early rheumatoid arthritis: A feasibility trial. Musculoskeletal Care. 2018 Mar;16(1):167-172. doi: 10.1002/msc.1214. Epub 2017 Oct 2. PMID 28967710
- [Background] van der Heijde D, Ramiro S, Landewe R, Baraliakos X, Van den Bosch F, Sepriano A, Regel A, Ciurea A, Dagfinrud H, Dougados M, van Gaalen F, Geher P, van der Horst-Bruinsma I, Inman RD, Jongkees M, Kiltz U, Kvien TK, Machado PM, Marzo-Ortega H, Molto A, Navarro-Compan V, Ozgocmen S, Pimentel-Santos FM, Reveille J, Rudwaleit M, Sieper J, Sampaio-Barros P, Wiek D, Braun J. 2016 update of the ASAS-EULAR management recommendations for axial spondyloarthritis. Ann Rheum Dis. 2017 Jun;76(6):978-991. doi: 10.1136/annrheumdis-2016-210770. Epub 2017 Jan 13. PMID 28087505
- [Background] Wendling D, Lukas C, Prati C, Claudepierre P, Gossec L, Goupille P, Hudry C, Miceli-Richard C, Molto A, Pham T, Saraux A, Dougados M. 2018 update of French Society for Rheumatology (SFR) recommendations about the everyday management of patients with spondyloarthritis. Joint Bone Spine. 2018 May;85(3):275-284. doi: 10.1016/j.jbspin.2018.01.006. Epub 2018 Mar 8. PMID 29407043
- [Background] Veldhuijzen van Zanten JJ, Rouse PC, Hale ED, Ntoumanis N, Metsios GS, Duda JL, Kitas GD. Perceived Barriers, Facilitators and Benefits for Regular Physical Activity and Exercise in Patients with Rheumatoid Arthritis: A Review of the Literature. Sports Med. 2015 Oct;45(10):1401-12. doi: 10.1007/s40279-015-0363-2. PMID 26219268
- [Background] Fongen C, Sveaas SH, Dagfinrud H. Barriers and Facilitators for Being Physically Active in Patients with Ankylosing Spondylitis: A Cross-sectional Comparative Study. Musculoskeletal Care. 2015 Jun;13(2):76-83. doi: 10.1002/msc.1088. Epub 2014 Nov 5. PMID 25370164
- [Background] Larkin L, Gallagher S, Fraser A, Kennedy N. Community-based intervention to promote physical activity in rheumatoid arthritis (CIPPA-RA): a study protocol for a pilot randomised control trial. Rheumatol Int. 2017 Dec;37(12):2095-2103. doi: 10.1007/s00296-017-3850-y. Epub 2017 Oct 17. PMID 29043493
- [Background] Lotzke D, Ostermann T, Bussing A. Argentine tango in Parkinson disease--a systematic review and meta-analysis. BMC Neurol. 2015 Nov 5;15:226. doi: 10.1186/s12883-015-0484-0. PMID 26542475
- [Background] Cleland CL, Hunter RF, Kee F, Cupples ME, Sallis JF, Tully MA. Validity of the global physical activity questionnaire (GPAQ) in assessing levels and change in moderate-vigorous physical activity and sedentary behaviour. BMC Public Health. 2014 Dec 10;14:1255. doi: 10.1186/1471-2458-14-1255. PMID 25492375